CLINICAL TRIAL: NCT04522895
Title: IDH2-Post-Allo-Trial: Enasidenib As Consolidation or Salvage Therapy for Patients with IDH2 Mutated AML or MDS Following Allogeneic Blood Stem Cell Transplantation
Brief Title: IDH2-Post-Allo-Trial for Patients with IDH2-mut Myeloid Neoplasms After Allo-SCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Celgene Corporation (Industry); Koordinierungszentrum für Klinische Studien Düsseldorf (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AG-221CL-AML-PI13299; 2019-001416-30 (EudraCT Number)
Record Dates: First submitted 2020-05-29; First posted 2020-08-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-12

CONDITIONS: Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Chronic Myelomonocytic Leukemia; IDH2 Gene Mutation; IDH2 R172; IDH2 R140
Keywords: IDH2 Gene Mutation; MDS; CMML; AML; allogeneic blood stem cell transplantation; maintenance; consolidation
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic | interventions — enasidenib

STUDY DESIGN:
Intervention Model Description: single arm
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Consolidation Arm (Experimental): Enasidenib (investigational product) will be started on day 1 for 28 days every 28 days for a maximum of 12 cycles. The starting dose of Enasidenib will be 100 mg once daily in every patient and may be reduced individually according to a dose modification scheme.
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — Participants receive up to 12 cycles of Enasidenib.

SUMMARY:
This is a prospective, open label, single arm, multi-centre phase II trial aiming to evaluate the safety and efficacy of Enasidenib (investigational product) as prophylactic consolidation in patients with IDH2-mutated MDS, CMML and AML in remission after allo-SCT.

DETAILED DESCRIPTION:
This is a prospective, open label, single arm, multi-centre phase II trial aiming to evaluate the safety and efficacy of Enasidenib (investigational product) as prophylactic consolidation in patients with IDH2-mutated MDS, CMML and AML in remission after allo-SCT.

Study Design:

* interventional
* prospective, open-label, single arm, multicenter phase-II trial
* total patients sample size: 50 patients
* number of trial sites: 11 all located in Germany and members of the EBMT

Patients with AML, MDS and CMML, in whom an IDH2 mutation has been detected at diagnosis prior allo-SCT, are eligible for consolidation therapy, if they are in complete hematological remission after first allo-SCT. IDH2 mutation might be absent at this time (CRMRDnegative), or might be detectable at submicroscopical levels (CRMRDpositive) given the high sensitivity of detection methods nowadays available. Remission will be evaluated within a screening period between day +25 and day +35. Evaluation of remission will be performed locally with IDH2 mutation analysis performed at an experienced local laboratory of the respective center. The report about IDH2 mutation testing at diagnosis has to be sent to the principle investigator for review at screening to include the patient; a BM sample will be stored for central retesting, which will be performed in batch during the course of the study. Having a documented hematological CR, patients will enter the treatment phase within 30 days after this BM evaluation (latest time point day +65) and start treatment with Enasidenib. They are envisaged to receive Enasidenib (100 mg per day, day 1-28) for up to 12 cycles (=12 months). Patients will go off protocol prematurely in case of relapse, intolerability of study treatment and in case of withdrawal of consent. In those patients who relapse during study treatment subsequent therapy for relapse will be performed according to the choice of the individual treating physician. Patients who finish study as planned or prematurely will be regularly followed for one year, lost to follow up, death or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

* Patients with myeloid malignancy (AML, MDS and CMML) and known IDH2 mutation (IDH2 R172 or R140 mutation) at diagnosis prior to first allo-SCT
* hematological CR after allo-SCT determined during screening period between day +25 and day +35 (the hematological remission will be confirmed locally by cytomorphological/histological evaluation)
* Hematopoietic recovery after transplantation indicated by an absolute neutrophil count of at least 1.000/µl and platelet count of at least 50.000/µl
* no previous therapy with Enasidenib or any other IDH2 inhibitor
* ECOG performance status ≤ 2 at study entry (s. Appendix)
* no active, steroid refractory GvHD treated with additional systemic immunosuppression within 4 weeks before inclusion
* no uncontrolled infection at inclusion
* Understand and voluntarily sign an informed consent form.
* Age ≥18 years at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements.
* Female of childbearing potential (FCBP) must:

Understand that Enasidenib can cause embryo-fetal harm when administered to a pregnant woman Agree to have a medically supervised pregnancy test within 72 hours prior study start and at day 1 of every treatment cycle Use effective contraception during treatment with Enasidenib and for at least 2 months after the last dose Coadministration of Enasidenib may increase or decrease the concentrations of combined hormonal contraceptives Avoid becoming pregnant while receiving Enasidenib Notify her study doctor immediately if there is a risk of pregnancy Agree to abstain from breastfeeding during study participation and for at least 30 days after study drug discontinuation Understand that Enasidenib may impair fertility in females of reproductive potential and this effect may be not reversible

- Males must: Understand that Enasidenib can cause embryo-fetal harm Use effective contraception during treatment with Enasidenib and for at least 2 months after the last dose of Enasidenib if engaged in sexual activity with a pregnant female or a female with childbearing potential Agree to notify the investigator immediately, if pregnancy or a positive pregnancy test occurs in his partner during study participation Understand that Enasidenib may impair fertility in males of reproductive potential and this effect may be not reversible

Exclusion Criteria:

* Any evidence of hematological relapse of the underlying IDH2-mutated myeloid malignancy (AML, MDS and CMML) determined during screening period until start of treatment
* Any previous prophylactic therapy given within the interval between allo-SCT and screening period
* Patients with myeloid malignancy (AML, MDS and CMML) and known IDH2 mutation (IDH2 R172 or R140 mutation) after second allo-SCT
* Active, steroid refractory GvHD treated with additional systemic immunosuppression within the last 4 weeks
* Uncontrolled infection
* Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
* Pregnant or lactating females
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Impaired renal function (GFR < 30 ml/min)
* Impaired hepatic function, as follows:

Aspartate aminotransferase (19) ≥3 x ULN or Alanine aminotransferase (ALT) ≥3 x ULN or Total bilirubin ≥3 x ULN or Alkaline Phosphatase ≥3 x ULN

* Known hypersensitivity to Enasidenib or any other component of the treatment
* Prior history of malignancy other than AML, MDS or CMML (except basal and squamous cell carcinoma or carcinoma in situ of the cervix or breast) unless the subject has been free of disease for ≥3 years
* Concurrent use of other anti-cancer agents or treatments
* Known positive for HIV or active infectious hepatitis, type A, B or C
* Participation in another study with ongoing use of unlicensed investigational product from 28 days before study enrollment until the end of the study (in cases where the investigational product has an unusually long half-life (e.g. antibodies), the interval until study enrollment must be at least five times the plasma half-life of the investigational product)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-08-27 (Actual); Primary Completion 2024-07-24 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Type, incidence and severity of adverse events specifying seriousness and expectedness (AE, SAE, SUSAR) | through study completion, an average of 2 years
  Number of participants with Adverse Events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Number of participants who maintain remission (molecular/hematological) after allo-SCT | through study completion, an average of 2 years
  Number of participants who maintain Remission (molecular/hematological) as a measure of efficacy
Overall Survival | through study completion, an average of 2 years
  Days from start of Treatment and from date of allo-SCT until death or last follow up as a measure of efficacy
Relapse-free Survival | through study completion, an average of 2 years
  Days from evaluation of remission at screening and from date of allo-SCT until relapse, death, or last follow up as a measure of efficacy
Non-relapse mortality | through study completion, an average of 2 years
  Days from evaluation of remission at screening and from date of allo-SCT until death without relapse or last follow up as a measure of efficacy
Relapse incidence | through study completion, an average of 2 years
  number of participants that relapse during the study as a measure of efficacy
Numbers of Participants Meeting Criteria of Treatment Failure | through study completion, an average of 2 years
  Number of participants who require any cellular or pharmacological intervention due to pending or frank relapse (defined as treatment-failure) as a measure of efficacy
Correlation of cytogenetics/molecular alterations and relapse-free survival | through study completion, an average of 2 years
  Comparison of relapse-free survival between different cytogenetics/molecular subtypes as a measure of efficacy using time to event curves and log-rank test
Incidence, course and severity of aGvHD and cGvHD | through study completion, an average of 2 years
  Incidence, course and severity of aGvHD and cGvHD as a measure of safety
Number of hospitalizations | through treatment completion, an average of 1 year
  Number of hospitalizations per participant as a measure of safety
Number of participants who require dose reductions for toxicity reasons | through treatment completion, an average of 1 year
  Number of participants who require dose reductions for toxicity reasons as a measure of safety
Number of participants who have to stop consolidation therapy due to toxicity (Consolidation Arm) | through treatment completion, an average of 1 year
  Number of participants who have to stop consolidation therapy due to toxicity as a measure of safety (Consolidation Arm)
Number of participants who can receive all 12 cycles of consolidation therapy(Consolidation Arm) | through treatment completion, an average of 1 year
  Number of participants who can receive all 12 cycles of consolidation therapy as a measure of Safety (Consolidation Arm)
Number of screened participants that can start consolidation therapy within the envisaged time frame (Consolidation Arm) | up to 65 days
  Number of screened participants that can start consolidation therapy within the envisaged time Frame as a measure of safety (Consolidation Arm)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Schroeder, PD Dr., Principal Investigator — University Hospital Duesseldorf Dept. of Hematology, Oncology and Clinical Immunology
Locations (11):
- Germany (11):
  - University Hospital Duesseldorf Dept. of Hematology, Oncology and Clinical Immunology, Düsseldorf, North Rhine-Westphalia
  - Uniklinik RWTH Aachen Klinik für Hämatologie, Onkologie, Hämostaseologie und Stammzelltransplantation (Med. Klinik IV), Aachen
  - Universitätsklinikum Köln Klinik I für Innere Medizin, Cologne
  - Universitätsklinikum Carl Gustav Carus Medizinische Klinik und Poliklinik I, Dresden
  - Universitätsklinikum Essen Klinik für Hämatologie und Stammzelltransplantation, Essen
  - Universitätsklinikum Frankfurt Med. Klinik II, Frankfurt
  - Universitätsklinikum Hamburg-Eppendorf Interdisziplinäre Klinik für Stammzelltransplantation, Hamburg
  - Universitätsklinikum Heidelberg Innere Medizin V: Hämatologie, Onkologie und Rheumatologie, Heidelberg
  - Universitätsklinikum Leipzig Medizinische Klinik und Poliklinik I, Hämatologie und Zelltherapie, Leipzig
  - Klinikum rechts der Isar der TU München Klinik und Poliklinik für Innere Medizin III, Hämatologie und Onkologie, München
  - Universitätsklinikum Münster Medizinische Klinik A / KMT Zentrum, Münster

IPD SHARING:
Plan to Share IPD: No